CLINICAL TRIAL: NCT07165145
Title: MicroHealth Project: Human Trial A A Randomized Comparative Trial to Examine the Impact of Organically vs Conventionally Grown Crops on the Human Gut Microbiome and Health
Brief Title: Effect of Agricultural Practices on Crops, Gut Microbiome, and Human Health
Acronym: MITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, Prof., Dr., Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NL88508.018.24
Record Dates: First submitted 2025-06-24; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Obesity Prevention; Microbiome Analysis
Keywords: Microbiome; Agricultural Strategies; Fruits and Vegetables; Diet; Organic and Conventional; Biological; Prevention
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Intervention Model Description: Study design:
  Double-blind randomized dietary intervention study, parallel design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A) 11 MetSyn participants (Active Comparator): Organic Fruits and Vegetables
  Interventions: Dietary Supplement: Organic Fruits and Vegetables
- B) 11 MetSyn participants (Active Comparator): Conventional Fruits and Vegetables
  Interventions: Dietary Supplement: Conventional Fruits and Vegetables
- C) 11 Healthy participants (Active Comparator): Organic Fruits and Vegetables
  Interventions: Dietary Supplement: Organic Fruits and Vegetables
- D) Healthy participants (Active Comparator): Conventional Fruits and Vegetables
  Interventions: Dietary Supplement: Conventional Fruits and Vegetables

INTERVENTIONS:
Dietary Supplement: Organic Fruits and Vegetables — Dietary Intervention
  Arms: A) 11 MetSyn participants; C) 11 Healthy participants
Dietary Supplement: Conventional Fruits and Vegetables — Dietary Intervention
  Arms: B) 11 MetSyn participants; D) Healthy participants

SUMMARY:
The human gut microbiome plays a regulatory role in host health, and is involved in metabolic, immune, and neurological processes. Diet shapes the gut microbiome; by providing essential nutrients, which sustain the existing microorganisms and by introducing foodborne microbes that modulate its composition. Notably, the impact of microbes from fruit and vegetables on the gut microbiome is relatively unexplored. Differences in agricultural practices, organic vs conventional strategies, can lead to variations in nutritional content and associated microbial communities in and on crops, underscoring the potential for variations in cultivated crops to influence the human gut microbiome's composition and function. This study aims to explore how crop cultivation practices affect the composition and function of the human gut microbiome, ultimately influencing overall health.

DETAILED DESCRIPTION:
Objective:

The primary objective of this study is to investigate the effect of differentially cultivated crops (organic versus conventional) on cardiometabolic health outcomes, as reflected by measurements of glucose metabolism and its relation to the gut microbiome composition and function.

The secondary objectives are to assess the effect of differently grown crops on gut microbiome composition and function, plasma and fecal short-chain fatty acid levels, including quantification of pesticide residues and other contaminants in blood and faeces. Additionally, changes will be evaluated in metabolomics of the blood and breath volatile organic compounds (QuinTron), as well as alterations in weight, body composition.

Double-blind randomized dietary intervention study, parallel design. A total of 40 male and female volunteers will be recruited for this study, aged 18-45 years.

20 will have a normal BMI of 19-25 with no current medical conditions, while the remaining 20 will have a BMI of 28-40 with three components of Metabolic Syndrome, drug-naïve.

Participants will be assigned to one of two groups for 4 weeks of dietary intervention. One group will receive produce from conventional agriculture, while the other receives produce from organic agriculture, with a specific focus on differently grown fruits and vegetables.

Both groups will receive:

* A weekly full meal recipe kit (6 days/week) with ingredients and instructions on preparation
* A separate weekly box containing additional fruits and vegetables (6 days/week)

ELIGIBILITY:
Inclusion Criteria:

* 22 Healthy Volunteers : healthy Caucasian adults with a BMI < 25 kg/m^2 will be recruited with no medical conditions.
* 22 Metabolically Impaired Participants: Caucasian adults with a BMI ranging from 28 kg/m^2 to 40 kg/m^2 with three components of Metabolic Syndrome, drug-naïve:

  * Elevated waist circumference (WC): with men having WC > 102 cm (40 inches) and women having a WC > 88 cm (35 inches).
  * High Fasting Plasma Glucose (FPG): a fasting plasma glucose level 110 mg/dL (6.1 mmol/L)
  * High Fasting Plasma Insulin (FPI): A fasting insulin level ≥25 μU/mL (or >16.7 pmol/L)
  * HOMA-IR score of ≥2.5

Exclusion Criteria:

* Use of antibiotic in the past 3 months or currently taking them
* Past/ Currently following a vegan, strictly organic or vegetarian diet.
* History of severe food allergies or intolerances that would render it unsafe for them to consume any of the fruits and vegetables provided. Exclusion will be determined on a case-by-case basis by the investigator.
* Inability or unwillingness to collect stools.
* Presence of overt type 1 diabetes mellitus (T1DM) and/or type 2 diabetes.
* Use of medications for type 2 diabetes: metformin, statin, proton pump inhibitors (PPI), H2 blockers, pioglitazone, active GLP-1 receptor agonists (e.g., exenatide, liraglutide).
* Prior or planned bariatric surgery, history of cholecystectomy.
* History of cardiovascular disease, having a severe disease of the digestive tract, such as celiac disease, Crohn's disease, active ulcerative colitis.
* Surgery scheduled for the trial duration period.
* Pregnant or nursing women.
* Smoking or illicit drug use. Use of >5 units of alcohol daily on average.
* History of neurological/neurodegenerative disorders.
* Participation in another concomitant clinical trial.
* Not residing in the Netherlands during study period (Sept-Nov 2025)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-07-05 (Estimated)

PRIMARY OUTCOMES:
Time in Range | At Baseline, week 4 (End-of-intervention)
  The primary objective of this study is to investigate the effect of deferentially cultivated crops (organic versus conventional) on glucose levels. Measured by the difference in time in range between the groups between baseline, end-of-diet intervention

SECONDARY OUTCOMES:
Continuous glucose monitoring | Between Baseline (week-1) and End-of-intervention (week4)
  Changes in glycemic variability, time above range, time below range and hypoglycemic episodes
Gut microbiome | Every week from baseline (week -1) to follow-up (week 6)
  Gut microbiome analysis will include qualitative and quantitative assessment via 16S and whole-genome sequencing, differential abundance testing with DESeq2, strain-level tracking using InStrain, and PERMANOVA to evaluate temporal effects
Body Composition | Baseline, End-of-intervention (week 4), Follow-up (week 6)
  Body Impedance Analysis: Free fat mass (kg; %). Fat mass (kg; %). Rest Metabolic Rate (kcal/day).
Anthropometric measurements | Baseline, week 4 and follow-up (week 6)
  Weight will be measured in kilograms (kg). Height will be measured in meters (m). These two measurements will also be combined to calculate Body Mass Index (BMI), defined as weight in kilograms divided by height in meters squared (kg/m²)
Dietary Intake | Baseline (week -1), End-of-Intervention (week 4), follow-up (week 6)
  Recorded of 3 days with "Eetmeter"
HbA1c | Baseline, End-of-Intervention (week 4), follow-up (week 6)
  Millimoles of HbA1c per mole of hemoglobin (mmol/mol)
HOMA-IR | Baseline, End-of-Intervention (week 4), follow-up (week 6)
  (Fasting Insulin * Fasting Glucose) / Constant
Leukocyte (differentation) | Between Baseline and End-of-intervention (week4), follow-up (week 6)
  ×10 9 /L
CRP | Between Baseline and End-of-intervention (week4), follow-up (week 6)
  C-reactive protein (mg/L)
Physical Activity Questionnaire | Between Baseline (week-1), End-of-intervention (week4) and Follow-up (week 6)
  Physical Activity Questionnaire (SQUASH - Short Questionnaire to Assess Health-enhancing Physical Activity): Assesses weekly physical activity levels across commuting, household, leisure, and work/school activities. Scores are reported in MET-hours per week, with higher scores indicating greater physical activity. Range of activity levels: Low: <10 MET-hours/week, Moderate: 10-29 MET-hours/week, High: ≥30 MET-hours/week.
Breath Gas H₂ | Baseline, End-of-Intervention (week 4), follow-up (week 6)
  Breath test performed with the QuinTron analyzer, measuring hydrogen (H₂) concentration in parts per million (ppm) as an indicator of fermentation.
Breath Gas CH₄ | Baseline, End-of-Intervention (week 4), follow-up (week 6)
  Breath test conducted with the QuinTron analyzer to measure methane (CH₄) concentration, expressed in parts per million (ppm), as an indicator of fermentation.
Breath Gas CO₂ | Baseline, End-of-Intervention (week 4), follow-up (week 6)
  Breath test conducted with the QuinTron analyzer to measure carbon dioxide (CO₂) concentration, expressed as a percentage (%) as control marker

CONTACTS AND LOCATIONS:
Overall Officials: Max Nieuwdorp, Dr. Prof., Principal Investigator — Dept of Vascular Medicine, Amsterdam UMC - AMC; Hilde H.J. Herrema, PhD, Principal Investigator — Dept of Vascular Medicine, Amsterdam UMC - AMC
Locations (1):
- Amsterdam UMC, locatie AMC, Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No